CLINICAL TRIAL: NCT04335513
Title: Trial of Early Initiation of CGM-Guided Insulin Therapy in Stage 2 T1D
Acronym: TESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Colorado, Denver (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-1767
Record Dates: First submitted 2020-03-17; First posted 2020-04-06 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Type 1 Diabetes; Prediabetic State; Dysglycemia; Autoimmune Diabetes
Keywords: Islet autoimmunity
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Early diabetes management and education including focused education based on pathophysiology of type 1 diabetes, factors which impact blood glucose, and effects of insulin using data from continuous glucose monitoring device (CGM) worn unblinded at least 20 days per month with interpretation and education on results. Early initiation of insulin therapy, when warranted based on a pattern of prolonged or repeated high blood glucose values.
  Interventions: Other: Early CGM-guided education and initiation of insulin therapy.
- Control (Active Comparator): Usual education and advice on glycemic surveillance based on protocols of TEDDY/DAISY/ASK (ongoing studies at BDC). This includes: blood glucose checks 2-3 times per month, participant-led contact with study personnel when abnormalities are noted and transition to clinical care when criteria for clinical type 1 diabetes are met.
  Interventions: Other: Usual care: glucometer surveillance and basic education.

INTERVENTIONS:
Other: Early CGM-guided education and initiation of insulin therapy. — Careful monitoring of children progressing from stage 2 to stage 3 T1D using continuous glucose monitor (CGM) technology, staged education targeted to assist families in recognizing evolving dysglycemia, and addressing glycemic abnormalities with early initiation of insulin can substantially reduce the HbA1c and risk of DKA at diagnosis, thereby changing the trajectory of the disease course.
  Arms: Intervention
Other: Usual care: glucometer surveillance and basic education. — * Usual education and advice on glycemic surveillance based on protocols of TEDDY/DAISY/ASK.
  * Blinded CGM for 10 days every 3 months to collect data on glycemic profile with basic feedback regarding changes.
  Arms: Control

SUMMARY:
This protocol is an intervention study to determine the best education and monitoring strategy for children ages 2-20 years with pre-symptomatic type 1 diabetes (T1D) because there currently exists no clinical guidelines for management of these children in early-stage T1D. This study hypothesizes that the trajectory of T1D can be changed, substantially reducing HbA1c and risk of DKA at diagnosis, through (1) careful monitoring of children progressing from stage 2 to stage 3 T1D using continuous glucose monitor (CGM) technology, (2) staged education targeted to assist families in recognizing evolving dysglycemia, and (3) addressing glycemic abnormalities with early initiation of insulin.

DETAILED DESCRIPTION:
Specific Aims:

Perform randomized controlled trial of intensive follow-up of stage 2 T1D participants utilizing continuous glucose monitoring (CGM) technology and early education of families to guide early insulin therapy with the goals of:

maintaining HbA1c less than 7.0%. avoiding adverse outcomes: ER visits, hospitalizations, DKA and severe hypoglycemia improving diabetes knowledge through optimal planned education as opposed to 'a crash course' at unexpected diagnosis event.

evaluating patient/caregiver satisfaction with diabetes care received evaluating impact of activity on glycemic profile Collect longitudinal biomarkers of beta-cell stress and dysfunction in stage 2 T1D.

Use longitudinal CGM data combined with "gold-standard" OGTT and HbA1c measures to provide evidence for CGM-based diagnostic criteria for stage 2 and stage 3 T1D.

Perform cost-analysis of intensive follow up protocol.

ELIGIBILITY:
1. Individuals identified in stage 2 T1D through ongoing screening studies at the Barbara Davis Center (ASK, DAISY, TrialNet, and TEDDY) who have given permission to be contacted about study opportunities.
2. Presence of islet autoimmunity with high risk of progression:

   i. positive for multiple islet autoantibodies at 2 or more visits -OR- ii. positive for a single high-affinity islet autoantibody at 2 or more visits
3. Evidence of dysglycemia (Stage 2 T1D) using any one of the following criteria:

I. Americal Diabetes Association (ADA) criteria:

1. fasting plasma glucose 100-125 mg/dL
2. OR 2-hour OGTT plasma glucose of 140-199 mg/dL
3. OR A1c 5.7-6.4%
4. OR ≥10% increase in A1c from previous visit

II. Dysglycemia on OGTT (TrialNet Criteria):

a. glucose above 200 mg/dL on 30, 60 OR 90 minute values

III. Dysglycemia on CGM worn for at least 5 days:

1. ≥15% of values above 140 mg/dL
2. OR peaks ≥ 200 mg/dL on ≥2 days
3. OR average sensor glucose ≥120 mg/dL

IV. Dysglycemia on finger stick blood glucose:

1. Fasting BG above 110 mg/dL on 2 or more days
2. OR 2 hour post-meal BG above 150 mg/dL on ≥ 2 days
3. OR single random BG > 200 mg/dL

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-04-30 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Diabetes Knowledge from baseline to 6 month follow-up. | Baseline, 6 months
  35-item diabetes questionnaire with possible responses true/false/don't know. Total score is the number of correct answers out of 35, with more correct answers indicating higher knowledge. Change from baseline to 6-month follow-up will be compared between groups
Continuous glucose monitor (CGM) % time >140 mg/dL | Baseline and 3, 6, 9 and 12 months
  Data obtained for Dexcom G6 wear with at least 5 days of data at each time point. Continuous glucose monitor (CGM) % time >140 mg/dL will be analyzed using linear mixed models incorporating data from all 5 time points, with an interaction between group and time to test for differences in change in outcome over time. Contrast statements will be used to test for comparisons of intervention vs controls.

SECONDARY OUTCOMES:
Change in HbA1c | Baseline and 3, 6, 9 and 12 months
  HbA1c from baseline to 52 weeks, adjusted for baseline
% with HbA1c <7.0% | Baseline and 3, 6, 9 and 12 months
  Percentage of individuals in each group with HbA1c <7.0%
Continuous glucose monitor (CGM) % time in range 60-140 mg/dL | Baseline and 3, 6, 9 and 12 months
  Data obtained for Dexcom G6 wear with at least 5 days of data.
Continuous glucose monitor (CGM) mean sensor glucose level (mg/dL) | Baseline and 3, 6, 9 and 12 months
  Data obtained for Dexcom G6 wear with at least 5 days of data.
Continuous glucose monitor (CGM) standard deviation sensor glucose level (mg/dL) | Baseline and 3, 6, 9 and 12 months
  Data obtained for Dexcom G6 wear with at least 5 days of data.
Continuous glucose monitor (CGM) coefficient of variation sensor glucose level (mg/dL) | Baseline and 3, 6, 9 and 12 months
  Data obtained for Dexcom G6 wear with at least 5 days of data.
Change in Pediatric Quality of Life Inventory (PedsQL 4.0) score over time | Baseline and 3, 6, 9 and 12 months
  The PedsQL 4.0 measures health-related quality of life across the domains of Physical Functioning, Emotional Functioning, Social Functioning, and School Functioning.
  ThePedsQL has parallel forms for parents of children aged 2-4, 5-7, 8-12, and 13-18 years. The child version has parallel forms for children aged 5-7, 8-12, and 13-18. Responses to items use a 5-point Likert scale (0 = never a problem, 4 = almost always a problem). Items are reverse scored and transformed to a 0 to 100 scale with higher scores indicating better quality of life.
Change in C-peptide response to Oral Glucose Tolerance Test (OGTT) | Baseline, 6 months, 12 months
  C-peptide measurement during standard OGTT, Area under the curve (AUC)
Change in insulin response to Oral Glucose Tolerance Test (OGTT) | Baseline, 6 months, 12 months
  insulin measurement during standard OGTT, Area under the curve (AUC)
Diabetes attitude survey change over time | Baseline, 6 months, 12 months
  10 item survey, each item answered on a likert scale from 1-5: (1) strongly disagree to (5) strongly agree. Scoring is on 4 scales: (1) "Value of Tight Control", scored on 4-20 points with higher score indicating agreement with importance of control; (2) "Psychosocial Impact", scored on 2-10 points with higher score indicating agreement with high impact of diabetes on psychosocial factors; (3) "Patient Autonomy", scored on 2-10 points with higher score indicating agreement with value of autonomy; and (4) "Confidence", scored on 2-10 points with higher score indicating confidence in knowledge and skills.

OTHER OUTCOMES:
Activity Monitoring daily steps | Monthly for months 0, 1, 2, 3, 4, 5, and 6 of study
  Activity tracker average of steps per day from at least 5 days of data at each time point. Average daily steps will be analyzed using linear mixed models incorporating data from all seven time points, with an interaction between group and time to test for differences in change in outcome over time. Contrast statements will be used to test for comparisons of interest (intervention vs controls).
Parental anxiety regarding diabetes risk | Baseline, 6 and 12 months
  Items from a questionnaire to study the psychological impact of diabetes risk. A 6-item short form of the state portion of the State-Trait Anxiety Inventory (STAI) will be used to assess parent anxiety about the child's diabetes risk at a single point in time. For example, parents were asked how often they feel "worried" specifically when they think about their child's risk of developing diabetes. Responses were scored on a 4-point scale and the 6-item score was then converted to a total score comparable to the 20-item State Anxiety Inventory score. Parents with STAI scores > 40 were considered to be highly anxious. STAI scores will be analyzed using linear mixed models incorporating data from all three time points, with an interaction between group and time to test for differences in change in outcome over time. Contrast statements will be used to test for comparisons of intervention vs controls.
Parental depression symptoms. | Baseline, 6 and 12 months
  Items from a questionnaire to study the psychological impact of diabetes risk. A 6-item set of questions quering frequency of depressive symptoms will be used to assess parent depressive symptoms at a single point in time. For example, parents will be asked about frequency of crying spells on a 4 point scale from (1) Not at all to (4) All of the time. Responses are scored from 6 to 24, with higher score indicating increased depressive symptoms.
Parental perception of ability to impact diabetes risk. | Baseline, 6 and 12 months
  Items from a questionnaire to study the psychological impact of diabetes risk. A 3 item survey, each item answered on a likert scale from 1-5: (1) strongly agree to (5) strongly disagree. Risk modification belief scoring is scored on 3-15 points with higher score indicating perception that risk of diabetes can be modified. Risk modification scores will be analyzed using linear mixed models incorporating data from all three time points, with an interaction between group and time to test for differences in change in outcome over time. Contrast statements will be used to test for comparisons of intervention vs control
Accuracy of parental risk perception. | Baseline, 6 and 12 months
  Items from a questionnaire to study the psychological impact of diabetes risk. The accuracy of parental perception of the child's risk for developing type 1 diabetes (T1D) is scored as accurate or inaccurate on a questionnaire (accurate: indicating the child's T1D risk was higher or much higher than other children's T1D risk; inaccurate: indicating the child's T1D risk was the same, somewhat lower or much lower than other children's T1D risk).
Parental worry regarding diabetes risk. | Baseline, 6 and 12 months
  Item from a questionnaire to study the psychological impact of diabetes risk. The frequency of worry regarding whether the child will develop diabetes is scored on a five item scale from (1) Never to (5) Very often. A score of 5 indicates increased level of worry.
Change in height over time | Baseline and 3, 6, 9 and 12 months
  Change in z-score of height, using CDC (Centers for Disease Control) standards for gender and age.
Change in weight over time | Baseline and 3, 6, 9 and 12 months
  Change in z-score of weight, using CDC standards for gender and age.
Change in BMI over time | Baseline and 3, 6, 9 and 12 months
  Change in z-score of BMI using CDC standards for gender and age.
Change in body fat over time | Baseline and 3, 6, 9 and 12 months
  Change in body fat percentile using Tanita bioelectrical impedance scale
Presence of one or more islet cell autoantibodies:over time | Baseline and 3, 6, 9 and 12 months
  islet autoantibodies measured in the blood: GAD65 autoantibody (GADA), islet antigen 2 autoantibody (IA-2A), insulin autoantibody (IAA), and zinc transporter 8 autoantibody (ZnT8A)
Change in glucose tolerance over time by Oral Glucose Tolerance Test (OGTT) | Baseline, 6 months, 12 months
  Abnormal glucose tolerance is defined as:
  Fasting plasma glucose ≥ 110 mg/dL (6.1 mmol/L) and < 126 mg/dL (7 mmol/L), or 2 hour plasma glucose ≥ 140 mg/dL (7.8 mmol/L) and < 200 (11.1 mmol/L), or 30, 60, 90 minute plasma glucose during OGTT ≥ 200 mg/dL (11.1 mmol/L)
  OGTT values diagnostic of diabetes is defined as:
  Fasting plasma glucose >126 mg/dL (7 mmol/L), or 2 hour plasma glucose >200 (11.1 mmol/L),
Continuous glucose monitor (CGM) % time <60 mg/dL | Baseline and 3, 6, 9 and 12 months
  Data obtained for Dexcom G6 wear with at least 5 days of data.
areal bone mineral density of the spine measured by osteodensitometry (DXA) | 3 and 9 month visits
  Measured in g/cm2 by Dual-energy X-ray absorptiometry (DXA)
areal bone mineral density of the proximal femur measured by osteodensitometry (DXA) | 3 and 9 month visits
  Measured in g/cm2 by Dual-energy X-ray absorptiometry (DXA)
Change in glycemic control over time | Baseline and 3, 6, 9 and 12 months
  1,5 anhydroglucitol
Insulin requirements | Baseline and 3, 6, 9 and 12 months
  total, basal and bolus insulin dose (Units/kg/day), both arms
Severe hypoglycemic episodes | 12 months
  frequency of severe hypoglycemic episodes (BG < 54 mg/dL)
diabetic ketoacidosis (DKA) episodes | 12 months
  frequency of DKA
ER visits and hospitalizations related to glycemia | 12 months
  frequency of ER/Hospitalizations
Adverse events | 12 months
  number, nature and severity of other adverse events
Assessment of frequency of use of CGM (continuous glucose monitor) system | 12 months
  Number of days using CGM
Change in Diabetes Knowledge from 6 month to 12 months follow-up. | 6 months to 12 months follow-up
  35-item diabetes questionnaire with possible responses true/false/don't know. Total score is the number of correct answers out of 35, with more correct answers indicating higher knowledge. Durability of knowledge from 6-month follow-up to 12 month follow-up will be compared between groups

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte I Frohnert, MD, PhD, Principal Investigator — Barbara Davis Center for Diabetes, University of Colorado
Locations (1):
- Barbara Davis Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No